CLINICAL TRIAL: NCT01367691
Title: Cardiac MR (CMR) in Cardiac Resynchronization Therapy (CRT) Non-responders: Therapy Optimization by Means of Tissue Characterization, Hemodynamic Analysis and Analysis of Myocardial Activation
Brief Title: Cardiac MR (CMR) in Cardiac Resynchronization Therapy Non-responders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Claas P. Naehle, Assistant Professor of Radiology, University Hospital, Bonn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206/10
Record Dates: First submitted 2011-06-01; First posted 2011-06-07 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Heart Failure
Keywords: CRT; heart failure; CMR; safety
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CRT reprogramming (Medtronic CRT) — CRT devices will be reprogrammed according to CMR analysis
  Other Names: Medtronic CRT devices by Medtronic are eligable to be included in this study.

SUMMARY:
Cardiac MR (CMR) will be used to assess myocardial activation and hemodynamics in patients with CRT.

Goals are to demonstrate that

* differences in Left ventricle (LV)- right ventricle (RV) pacing delays cause differences in myocardial activation
* differences in LV-RV pacing delays cause differences in LV/RV hemodynamics

and to use these data to optimize CRT.

DETAILED DESCRIPTION:
CMR will be performed in patients under CRT who are currently not responding to CRT. Different LV-RV delays will be programmed during CMR and LV function and different dyssynchrony parameters will be assessed. Results will be used to determine the optimal LV-RV delay, and CRT-devices will be reprogrammed accordingly. Improvement in NYHA-class/conversion to therapy responder will be determined clinically after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* presence of CRT device
* CRT non responder

Exclusion Criteria:

* pregnancy
* end-stage renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
improvement in NYHA-class | 6 months

SECONDARY OUTCOMES:
safety of CMR in CRT-patients | 6 months
  pacing capture threshold, sensing and lead impedances will be monitored for significant and/or clinically relevant changes.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, University of Bonn, Bonn, North Rhine-Westphalia, Germany